CLINICAL TRIAL: NCT04040036
Title: Effects of Virtual Reality on Pain, Fear and Anxiety During Blood Draw in Children Aged 5-12 Years Old: A Randomized Controlled Study
Brief Title: Effects of Virtual Reality on Pain, Fear and Anxiety During Blood Draw in Children Aged 5-12 Years Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Asistant Professor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0000-0002-2229-616X
Record Dates: First submitted 2019-06-27; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Pain; Anxiety State; Fear; Child, Only
Keywords: blood draw
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: prospective, parallel trial design
Who Masked: Participant
Masking Description: Children Aged 5-12 Years Old
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR-Rollercoaster (Experimental): The children in the VR groups were told to watch the video by wearing virtual glasses during the blood draw. By wearing the VR headsets in the VR-Rollercoaster Group, individuals feel as if they are getting on and riding a rollercoaster. The rollercoaster speeds up and slows down.
  Interventions: Behavioral: Children watch applications by wearing the virtual headset during the blood draw.
- VR-Ocean Rift (Experimental): The children in the VR groups were told to watch the video by wearing virtual glasses during the blood draw. By wearing the VR headsets in the VR-Ocean Rift Group, individuals can take an underwater tour with 12 different marine animals with slow music.
  Interventions: Behavioral: Children watch applications by wearing the virtual headset during the blood draw.
- Control (No Intervention): They would be monitored during the procedure if their informed consent was received. Control group children did not receive any distraction techniques.

INTERVENTIONS:
Behavioral: Children watch applications by wearing the virtual headset during the blood draw. — wearing the virtual headset
  Arms: VR-Ocean Rift; VR-Rollercoaster

SUMMARY:
Virtual Reality (VR) has firmly stood amongst other technological devices and can easily be adapted to clinical procedures due to its low cost. It can be easily used particularly in pediatric care units because it appeals to various age groups and can be adapted to mobile phones. Virtual Reality (VR) can be used during painful procedures in children. The aim of this study was to evaluate the effects of two different VR methods on procedure-related pain, fear and anxiety of children aged 5-12 years old during blood draw. This randomized controlled study used parallel trial design.

DETAILED DESCRIPTION:
Aim and Hypothesis

The aim of this study was to evaluate the effects of two different VR methods on procedure-related pain, fear and anxiety levels of children aged 5-12 years old during blood draw. The hypotheses of this study were to:

H1: Children in the two different VR groups will have significantly less procedure-related pain than those in the control group.

H2: Fear and anxiety scores of the children in the two different VR groups will be reduced than those in the control group.

Study sample This prospective, randomized controlled study was conducted at a university hospital special blood draw unit in Izmir, Turkey between September 2017 and November 2017. A parallel trial design was used describing two different VR groups (VR-Rollercoaster group and VR-Ocean Rift group) and a control group (no VR device used) as the third arm. Children aged 5-12-year-old who underwent blood draw were eligible to participate (n=136). This age group was selected because they were open to co-operation and more curious about technology.

It was determined that 18 children in pain dimension and 19 children in fear dimension should be sampled in each group according to the one-way analysis of variance for the comparison of mean self-reported pain and fear scores (Canbulat et al., 2014), based on a power of .95 and an acceptable Type I error size of .05 in three groups in the Gpower 3.1.0 statistical program. It is planned that each group will consist of 45 children, considering that the parametric test assumptions can be fulfilled and lost in the study.

Randomization One hundred seventy-three children were assessed for eligibility; 32 children were excluded; refused to participate (n = 18); had chronic or genetic diseases (n = 12); had visual problem (n = 2). One hundred forty-one children randomized; 5 children were excluded/incomplete data collection (wanted to remove VR during the procedure). The final sample comprised 136 children (Figure 1) (Schulz, Altman, Moher, & the CONSORT Group, 2010).

The children meeting the inclusion criteria's were included in the study; (a) aged 5-12-year-old, (b) underwent blood draw, (c) had no chronic or genetic diseases, (d) had no visual problem or eyeglasses. The informed consent was received form children and parents. Their sample characteristics recorded. They were allocated by the blocked randomization; gender (2 blocks) and age groups (5-8 / 9-12-year-old: 2 blocks). The allocation concealment was guaranteed by a computer-generated number table by the researcher. Children and parents did not know which group they were included at the time of allocation concealment.

Instruments Demographic Form. This form included the child's gender, age, the last blood draw time, blood draw success and also the parent demographics such as age, educational level.

Wong-Baker FACES (WB-FACES) Pain Rating Scale. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10.

The Child Fear Scale (CFS). This scale is a one-item self-report measure for measuring pain-related fear in children. It ranges from a no fear (neutral) face on the far left to a face showing extreme fear on the far right. The rater responds indicates the level of fear for children aged 5-10 years (McMurtry, Noel, Chambers, & McGrath, 2011).

The Children's Anxiety Meter (CAM). It assesses children's anxiety in clinical settings and uses before medical procedures. Children are asked to mark how he/she feel "right now" to measure state anxiety (CAM-S). (Kleiber & Mccarthy, 2006). Scores range from 0 to 10. It validated at children aged 4-10 years during an intravenous procedure.

Data collection A single researcher (called Z) gave information about the study to the participants in the waiting area in the entrance of a private blood draw unit. The informed consent was received form children and parents. Their sample characteristics recorded. The allocation concealment was guaranteed by a computer-generated number table by the researcher Z. Children and parents did not know which group they were included at the time of allocation concealment. The researcher Z informed the researcher G that children allocated to which group.

CFS and CAM-S were administered by another researcher (called D) to the children to assess their fear and anxiety levels about blood draw. The researcher D did not know which group children were included, was blinded to the groups. The children were told that their blood would be drawn, and that they would be asked to rate their fear and anxiety on CFS and CAM-S just before the blood draw. The instructions about the scales were read to the children. Children rated the score on the paper. Afterwards, the children's parent was asked to rate the CFS and CAM-S according to child's fear and anxiety. Child and parent were blind to each other score. Finally, the researcher D rated CFS and CAM-S. The researcher D was not blinded to the children and parent's score because she collected the scores. The children and their parents were taken into the unit where the blood draw was performed. All children were allowed to keep their family nearby during the blood draw.

Blood draw procedure; It was performed 5 pediatric nurse specialists in this special blood draw unit. There were 5 blood collection cabins in the unit, the child went to the cabin according to the sequence number. Each blood draw cabin had one nurse. When the child went to the cabin, the nurse asked for the name of the child and told the child to sit in the blood draw chair. His/her parent also sat in a chair next to the child. The nurse introduced the materials to be used in the blood draw process, asked the child which arm wants blood drawn. After allowing the child to blood draw, the nurse performed the procedure. If the procedure failed, the child was asked to allow the blood draw from the other arm. If the child did not want to blood draw immediately, it was expected for a while. The nurse performed the procedure again when the child is ready.

Scripted verbal protocol used for nurses. It was stated that children in the control group would not be administered a non-pharmacological method. The children in the VR groups were told to watch the video by wearing virtual glasses. However, it was not explained which VR group the child was. The nurses were blinded to the VR groups. They were told to stop the procedure if child wanted to remove the virtual glasses. The nurses were asked to rate the WB-FACES for all of the children after the blood draw. The nurses had no conﬂict of interest, all of them agreed to participate.

Control Group; The first researcher (called G) explained to the patients in the control group that no additional procedure would be performed and they would be monitored during the procedure if their informed consent was received. Control group children did not receive any distraction techniques.

The virtual headsets were introduced to the children in the intervention groups by the researcher G, and they were told that they could watch applications by wearing the virtual headset during the procedure. The VR applications were chosen by the researchers. Since fear and anxiety, as well as pain, were assessed in the present study, the researchers preferred one of the applications to be more remarkable/distractor and the other to be more relaxing. Before the study was conducted, 10 children aged between 5 and 12 years old were asked to watch these two applications, and no negative feedback was received. By wearing the VR headsets in the VR-Rollercoaster Group, individuals feel as if they are getting on and riding a rollercoaster. The rollercoaster speeds up and slows down. By wearing the VR headsets in the VR-Ocean Rift Group, individuals can take an underwater tour with 12 different marine animals with slow music.

The children were excluded from the study that they wanted to take off the virtual headset during the procedure. When the child wanted to take off the virtual headset, blood draw procedure was stopped and immediately the virtual headset was removed and blood draw procedure continued.

During the procedure, the researcher G monitored the children and recorded the procedure success at the same time. When the blood started to flow into the tube within 5 seconds with disposable Vacutainer®, the blood draw was considered successful.

After the procedure finished, the researcher G, the children and their parents went to the waiting area in the entrance of a private blood draw unit. The researcher G gave the children a pen and asked them to rate the fear and anxiety they experienced during the blood draw procedure on the CFS and CAM-S again and also asked to rate their pain levels on the WB-FACES. Afterwards, their parents were asked to rate the CFS, CAM-S and WB-FACES. The researcher G also rated CFS, CAM-S and WB-FACES. After the children left from the unit, the nurse who performed the procedure was asked to rate the WB-FACES. The nurse was blinded to the child, parent and researcher's score. The researcher G was not blinded because she collected the scores. The researcher G and researcher D were blinded to each other's scores. The researcher G didn't know the scores before the blood draw.

Ethics Ethical approval was received from the Non-Invasive Clinical Studies Ethics Committee of University (3481GOA 2017/20-02) and institutional permissions (71995408-000-10575). The researcher informed the children and their parents about the aim of the study and obtained written consent forms from parents.

Data Analysis Data analysis was conducted by the Researcher M, was blinded to the groups. Percentages and means were used to evaluate the sample demographics. The data were analyzed using SPSS (22.0) software. The normal distribution of the data was assessed by Kolmogorov-Smirnov and Shapiro-Wilk tests. Sample characteristics were compared with Chi Square test in the three groups. The pain scores of the different VR and control groups were not normally distributed, the comparison of the pain scores of the three groups were evaluated with Kruskal Wallis analysis. One-way ANOVA test was used to compare the mean scores of the groups because of the normal distribution of fear and anxiety scores of the three groups before and after the blood draw. For any statistically significant differences between the three groups, post hoc pairwise comparisons were conducted using the Bonferroni adjustment. The effect of three groups on predicting fear and anxiety, and the effect of decrease in fear and anxiety were evaluated with linear regression analysis. The data were analyzed by using Tolerance and VIF values. p values were accepted as statistically significant <.05.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-12-year-old who underwent blood draw procedure were eligible to participate in this study.

Exclusion Criteria:

Participants were excluded from the study if they were

* refused to participate
* had chronic or genetic diseases
* had visual problem.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Pain assesed by Wong-Baker FACES | an average of 3 months
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst). This scale was assessed using self-report and reports from the parents, the researcher and the nurse who attempted the blood draw after the blood draw procedure in this study.

SECONDARY OUTCOMES:
Procedure Related Fear | an average of 3 months
  The Child Fear Scale (CFS) used. This scale is a one-item self-report measure for measuring pain-related fear in children. This one-item scale consists of five sex-neutral faces. It ranges from a no fear (neutral) face on the far left to a face showing extreme fear on the far right. The rater responds indicates the level of fear. It can be used by the parents and researchers before and during the procedure for children aged 5-10 years.CFS were administered by the researcher to the children to assess their fear levels about blood draw before and after blood draw procedure.
Procedure Related Anxiety | an average of 3 months
  The Children's Anxiety Meter (CAM) used. It assesses children's anxiety in clinical settings and uses before medical procedures. The CAM is drawn like a thermometer with a bulb at the bottom, also includes horizontal lines at intervals going up to the top. Children are asked to mark how he/she feel "right now" to measure state anxiety (CAM-S). (Kleiber & Mccarthy, 2006). Scores range from 0 to 10. It validated at children aged 4-10 years during an intravenous procedure.CAM were administered by the researcher to the children to assess their anxiety levels about blood draw before and after the blood draw procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, Study Director — Dokuz Eylul University Nursing Faculty Pediatric Nursing Department
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No